CLINICAL TRIAL: NCT02743247
Title: Identification of Drug-drug Interaction Between Tacrolimus and Mycophenolate Mofetil in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Yon Su Kim, Principal Investigator, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 17-2015-006-4
Record Dates: First submitted 2015-12-18; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteer
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus and Mycophenolate mofetil (Experimental): Tacrolimus 5mg single dose, Mycophenolate 1,000mg single dose, Tacrolimus 5mg and Mycophenolate 1,000mg single dose.
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Tacrolimus
  Other Names: Prograf
Drug: Mycophenolate mofetil
  Other Names: Cellcept

SUMMARY:
Coadministration of tacrolimus and mycophenolate mofetil is frequent in kidney transplantation. Due to narrow therapeutic range of tacrolimus and mycophenolate mofetil, therapeutic drug monitoring with dose adjustment is required. Investigating pharmacokinetic interplay between two drugs enables fine dose adjustment, while mechanism of drug interaction between two drugs is still not well understood. Therefore, an open-label, three period, single dose trial is planned to investigate the drug interaction between tacrolimus and mycophenolate mofetil.

DETAILED DESCRIPTION:
Study consists of three periods with fixed sequence: 1) single dose of mycophenolate mofetil 1,000mg; 2) single dose of tacrolimus 5mg; 3) single dose of mycophenolate mofetil 1,000mg and tacrolimus 5mg. All subjects have one week of washing period between single dose administration. Blood samples are drawn up to 72 hours after drug administration. Single nucleotide polymorphisms known to result in pharmacokinetic variability of study drug are also investigated. Drug interaction is going to be assessed through the ratio of area under the concentration curve of one drug in the presence or absence of another drug.

ELIGIBILITY:
Inclusion Criteria:

* Male adult with age of 19-45
* Weight difference between ideal and actual body weight is less than 20%
* Previous healthy with no known disease
* Considered normal on physical exam, clinical laboratory tests(complete blood count, electrolyte, renal and hepatic function) and electrocardiogram
* Never been heavy-drinker within one month prior to trial initiation and able to abstain from alcohol during trial

Exclusion Criteria:

* Ever smoked within one year prior to trial initiation
* Took other drugs (including herbal medicine) within one month prior to trial initiation
* Alcohol or drug abuser
* Participated another clinical trial within three months
* Considered inadequate under investigator's discretion

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve (AUC) of Tacrolimus and Mycophenolate mofetil | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours post-dose

SECONDARY OUTCOMES:
Peak Concentration of Tacrolimus and Mycophenolate mofetil | 0, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours post-dose
Adverse Drug Reaction | through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Yon Su Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea